CLINICAL TRIAL: NCT02859922
Title: A Comparison Between the Supreme Laryngeal Mask Airway and the Laryngeal Tube Suction During Spontaneous Ventilation: A Randomized Prospective Study
Brief Title: Comparison Between the Supreme Laryngeal Mask Airway and the Laryngeal Tube Suction During Spontaneous Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: BnaiZionMC-16-LG-002
Record Dates: First submitted 2016-07-25; First posted 2016-08-09 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Laryngeal Tube Supreme Spontaneous Ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supreme Laryngeal Mask Airway (Active Comparator): Supreme Laryngeal Mask Airway
  Interventions: Device: Supreme Laryngeal Mask Airway
- Laryngeal Tube Suction Disposable (Active Comparator): Laryngeal Tube Suction Disposable
  Interventions: Device: Laryngeal Tube Suction Disposable

INTERVENTIONS:
Device: Laryngeal Tube Suction Disposable — Laryngeal Tube Suction Disposable
  Arms: Laryngeal Tube Suction Disposable
Device: Supreme Laryngeal Mask Airway — Supreme Laryngeal Mask Airway
  Arms: Supreme Laryngeal Mask Airway

SUMMARY:
The study compared the Laryngeal Tube Suction (LTS-D) Disposable with the Supreme Laryngeal Mask Airway (SLMA) during spontaneous ventilation. The investigators hypothesized that the LTS-D and the SLMA perform similarly during spontaneous ventilation despite differences in their structural design.

DETAILED DESCRIPTION:
The Supreme Laryngeal Mask Airway (SLMA), (Intavent Orthofix, Maidenhead, UK), and Laryngeal Tube Suction -Disposable (LTS-D, (VBM Medizintechnik GmbH, Sulz, Germany), are second generation single-use supraglottic airway devices (SADs) with gastric access, for airway management in spontaneously and mechanically ventilated patients undergoing general anesthesia.

The SLMA has been compared to the Proseal Laryngeal Mask Airway (PLMA) during mechanical and spontaneous ventilation the LTS II (multiple use version of the LTS-D) with the PLMA.

Recently, the LTS-D and SLMA have been compared when used during pressure controlled mechanical ventilation.

To date, there is no published data comparing the SLMA to the LTS-D during spontaneous ventilation. The investigators hypothesized that the SLMA and LTS-D perform similarly during spontaneous ventilation despite differences in their structural design.

The chief aim of this prospective randomized study was to compare the SLMA and the LTS-D with respect to 1) Oxygen saturation and End Tidal carbone dioxide during spontaneous ventilation, 2) time to achieve an effective airway, 3) ease of insertion, 4) need for interventions to achieve an effective airway, 5) cuff seal (leak) pressure at an intracuff pressure of 60 cm H2O, 6) ventilatory variables during spontaneous ventilation, 7) fiberoptic score, 8) adverse perioperative events.

ELIGIBILITY:
Inclusion criteria:

* Patients, American Society of Anesthesiologists ( ASA) physical status I and II, with normal airways for minor elective surgery.

Exclusion Criteria:

* Age <18 years,
* Weight <50 kg,
* Cervical spine disease limiting neck a known difficult airway, and
* Patients with active gastroesophageal reflux.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation in percent | 30 min
  The data were recorded by the Anesthesia Delivery Unit (Datex-Ohmeda, Helsinki, Finland). monitor from starting the establishment of spontaneous ventilation until the device was removed

SECONDARY OUTCOMES:
Time to achieve an effective airway in sec | 15 sec
  The time was measured in seconds after the anesthesiologist removed the facemask and insert the device and the square-wave capnograph tracing was observed.Two attempts at insertion were permitted. If unsuccessful the patient's airway was managed with a conventional endotracheal tube.

OTHER OUTCOMES:
Sore throat in Numeric Rating Scale. | After the patient was released from Post Anesthesic Care Unit and 24 hours postoperatively.
  Sore throat was assessed subjectively by the patient using the 0-10 Numeric Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Gaitini, M.D., Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Luis A Gaitini M.D., Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes